CLINICAL TRIAL: NCT05563077
Title: Effects of Two Types of Aerobic Training on Ambulatory Blood Pressure in Hypertensives: a Systems Biology Approach
Brief Title: Aerobic Exercise and Resistant Hypertension
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Ruilope, Principal investigator, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UEM
Record Dates: First submitted 2022-09-21; First posted 2022-10-03 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Resistant Hypertension
Keywords: physical exercise; blood pressure; proteomics; resistant hypertension
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The sample of this study will be randomized in a 1:1:1 ratio (www.randomizer.org) based on a computer-generated random allocation sequence, and will be concealed using sequentially numbered, opaque, sealed envelopes to MIIT, MICT and control groups.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Care providers and outcomes assessors will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Moderate-intensity interval training (MIIT) (Experimental): 24 participants with resistant hypertension will perform moderate-intensity interval training.
  Interventions: Other: Moderate-intensity interval training (MIIT)
- Moderate-intensity continuous training (MICT) (Experimental): 24 participants with resistant hypertension will perform moderate-intensity continuous training.
  Interventions: Other: Moderate-intensity continuous training (MICT)
- Usual care (No Intervention): 24 participants with resistant hypertension will maintain usual care for 4 months.

INTERVENTIONS:
Other: Moderate-intensity interval training (MIIT) — MIIT group: participants will perform 3 sessions per week for 4 months. Each session will involve a ∼3 min warm-up (joint mobility exercises and walking at ∼2.2 METs), a ∼40-50 min main period (∼6-7 reps of 4 min at ∼4.2 METs, with 3 min of active recovery at ∼2.2 METs between each interval), and a ∼3-min cool-down (joint mobility exercises and walking at ∼2.2 METs). We will select the same aerobic dose of training (i.e., kcal/kg of body weight per week) to match total energy expenditure in both exercise groups.
  Arms: Moderate-intensity interval training (MIIT)
Other: Moderate-intensity continuous training (MICT) — MICT group: participants will perform 3 sessions per week for 4 months. Each session will involve a ∼3 min warm-up (joint mobility exercises and walking at ∼2.2 METs), a ∼40-50 min main period at ∼3.2 METs, and a ∼3-min cool-down (joint mobility exercises and walking at ∼2.2 METs).
  Arms: Moderate-intensity continuous training (MICT)

SUMMARY:
This study will examine the effects of 4 months of aerobic interval training versus continuous aerobic training on ambulatory blood pressure (ABP) and novel plasma protein biomarkers in patients with resistant hypertension. A randomized controlled trial will be performed including two exercise groups and a control group: a) moderate-intensity interval training (MIIT); b) moderate-intensity continuous training (MICT); c) usual care. MIIT could represent a superior training modality that exceeds the benefits of MICT in patients with resistant hypertension.

DETAILED DESCRIPTION:
Hypertension is associated with an increased risk of cardiovascular morbidity and mortality, and its high prevalence remains a worldwide concern. Ambulatory blood pressure monitoring (ABPM) is recognized in the diagnosis and management of hypertension, and can control blood pressure better than clinic assessment. Different studies have examined the effects of aerobic training on ABP in patients with hypertension, but the effects of moderate-intensity interval training (MIIT) and moderate-intensity continuous training (MICT) on ABP and novel plasma protein biomarkers that could potentially serve to identify cardiovascular risk, have not yet been examined in patients with resistant hypertension.To fill this gap, our aims are to determine the effects of MIIT and MICT for 4 months on ABP (primary endpoint), and on proteomic biomarkers (secondary endpoints) in patients with resistant hypertension. A total of 72 participants will be randomly divided into three groups: the first group (n=24) will perform MIIT, the second group (n=24) will perform MICT, and the third control group (n=24) will maintain usual care for 4 months. All will receive usual care for 4 months, with the structured physical exercise as the only relevant change in the intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with resistant hypertension (RH) (i.e., systolic BP/diastolic BP >130/80 mmHg according to the American College of Cardiology/American Heart Association) despite the concurrent use of three or more antihypertensive drugs - commonly including a diuretic, a long-acting calcium channel blocker, and a blocker of the renin-angiotensin system. RH also includes patients whose BP achieves target values on ≥ 4 antihypertensive. medications (i.e., 'controlled' RH).
* Adherence to prescribed medications.
* Willing to be randomized to one of the 3 groups.
* Informed consent.

Exclusion Criteria:

* Exclusion criteria will include exercising more than 30 minutes on 3 days or more weekly.
* Severe ischemic heart disease, major psychiatric disorder and other health contraindications that may interfere in the evaluations or interventions.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Change in 24-hour ambulatory blood pressure | Baseline to immediate post-treatment (4 months)
  Ambulatory SBP and DBP will be recorded with a validated oscillometric device over 24 hours.

SECONDARY OUTCOMES:
Change in plasma proteome | Baseline to immediate post-treatment (4 months)
  Olink's Proximity Extension Assay (PEA) technology, using the inflammation panel, will be used to evaluate changes in the plasma proteome.
Changes in albuminuria | Baseline to immediate post-treatment (4 months)
  Albuminuria will be determined from the albumin/creatinine ratio in urine.
Changes in glomerular filtration rate | Baseline to immediate post-treatment (4 months)
  The estimated glomerular filtration rate (eGFR) will be determined from serum creatinine levels using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.

OTHER OUTCOMES:
Change in aerobic capacity | Baseline to immediate post-treatment (4 months).
  VO2 will be measured breath-by-breath using a gas exchange analysis system.
Change in body composition | Baseline to immediate post-treatment (4 months)
  Dual-energy X-ray absorptiometry (DXA) scans will performed to measure body composition (fat mass and lean mass).
Change in lipid profiles | Baseline to immediate post-treatment (4 months).
  Blood analysis will be performed to evaluate HDL-C, LDL-C, total cholesterol, and triglyceride levels.
Change in echocardiography-determined left ventricular ejection fraction | Baseline to immediate post-treatment (4 months).
  The percentage of blood volume ejected from the left ventricle with each systolic contraction [(left ventricular end-diastolic volume - left-ventricular end-systolic volume)/ left ventricular end-diastolic volume] × 100.
Change in echocardiography-determined relative wall thickness (RWT) | Baseline to immediate post-treatment (4 months)
  The RWT will be calculated using the following formula:
  RWT = (Interventricular septum + left ventricular posterior wall thickness)/Left ventricular end-diastolic diameter).
Change in echocardiography-determined left ventricular global longitudinal strain (LV-GLS) | Baseline to immediate post-treatment (4 months)
  Two-dimensional speckle tracking echocardiography will be used to determine LV-GLS The Auto Strain function will be used for out-of-cart strain assessment on saved records. GLS values will be obtained by analyzing multi-camera perspectives, including two-, three- and four-camera views.
Change in echocardiography-determined left ventricular end-diastolic diameter (LVEDD) | Baseline to immediate post-treatment (4 months)
  LVEDD will be measured using two-dimensional guided M-mode imaging following recommendations from the American Society of Echocardiography.
Change in echocardiography-determined left ventricular (LV) mass | Baseline to immediate post-treatment (4 months)
  LV dimensions will be expressed relative to body surface area (in m x^2).
Change in echocardiography-determined left ventricular end- diastolic volume (LVEDV) | Baseline to immediate post-treatment (4 months)
  We will use the following equation to measure LVEDV:
  LVEDV (mL) = [7.0/(2.4 + Left ventricular end-diastolic diameter)] × Left ventricular end-diastolic diameter x^3.
Change in echocardiography-determined interventricular septal wall thickness (IVS) | Baseline to immediate post-treatment (4 months)
  IVS will be measured using two-dimensional guided M-mode imaging following recommendations from the American Society of Echocardiography.
Change in echocardiography-determined left ventricular posterior wall thickness (LVPW) (diastole) | Baseline to immediate post-treatment (4 months)
  LVPW will be measured using two-dimensional guided M-mode imaging following recommendations from the American Society of Echocardiography.
Change in carotid intima-media thickness (IMT) | Baseline to immediate post-treatment (4 months)
  The IMT will be measured in a long axis view in each distal common carotid artery, at least 5 mm proximal to the bifurcation, as the mean distance between the luminal-intimal and the medial-adventitial interfaces over a 10-mm length in the far wall.
Change in femoral intima-media thickness (IMT) | Baseline to immediate post-treatment (4 months)
  The IMT will be measured in a long axis view in each distal common carotid artery, at least 5 mm proximal to the bifurcation, as the mean distance between the luminal-intimal and the medial-adventitial interfaces over a 10-mm length in the far wall.
Change in carotid plaque maximal thickness | Baseline to immediate post-treatment (4 months)
  A plaque will be defined as the presence of a focal wall thickening ≥50% greater than the surrounding vessel wall, a focal region with an IMT measurement ≥1.5 mm, or a ≥0.5 cm protrusion into the lumen exceeding the IMT.
Change in femoral plaque maximal thickness | Baseline to immediate post-treatment (4 months)
  A plaque will be defined as the presence of a focal wall thickening ≥50% greater than the surrounding vessel wall, a focal region with an IMT measurement ≥1.5 mm, or a ≥0.5 cm protrusion into the lumen exceeding the IMT.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Ruilope, PhD, Principal Investigator — UEM
Locations (1):
- Universidad Europea Madrid (UEM), Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No